CLINICAL TRIAL: NCT00148538
Title: Type 1 Diabetes Aerobic and Resistance Exercise (T1-DARE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GA-3-05-1903-RS
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; Resistance Exercise; Aerobic Exercise; Exercise & Disease; Exercise; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): resistance exercise
  Interventions: Behavioral: Resistance and/or Aerobic Exercise
- 2 (Active Comparator): Aerobic and Resistance exercise
  Interventions: Behavioral: Resistance and/or Aerobic Exercise

INTERVENTIONS:
Behavioral: Resistance and/or Aerobic Exercise — Resistance and/or Aerobic Exercise
  Other Names: non applicable

SUMMARY:
This is a randomized controlled trial evaluating different exercise modalities in previously inactive subjects with type 1 diabetes.

The primary objective of this study is to determine the effects of resistance exercise training, and of aerobic exercise training, on glycemic control (A1c) in previously inactive individuals with type 1 diabetes, with background therapy meeting modern standards, including multiple daily insulin injections or insulin pump, carbohydrate counting, frequent glucose monitoring, and utilization of glucose monitoring to adjust CHO and insulin for exercise.

Secondary aims: In type 1 diabetic individuals receiving therapy meeting the criteria above, to determine the effects of resistance exercise training and aerobic exercise training on frequency of hypoglycemia, body composition, lipids, C-reactive protein and quality of life.

Hypotheses:

1. Subjects randomized to resistance exercise (R and AR combined) will have greater reductions in A1c than in those not randomized to resistance exercise (A and C combined).
2. Subjects randomized to aerobic exercise (A and AR combined) will show a trend to greater HbA1c reduction than those not randomized to aerobic exercise (R and C combined).

Secondary hypotheses: We expect that both aerobic and resistance exercise will show trends to improvement in most listed secondary outcomes.

DETAILED DESCRIPTION:
Background: Type 1 diabetes is characterized by complete or near-complete absence of insulin secretion, generally due to autoimmune disease. Cardiovascular disease (CVD) risk in type 1 diabetes is just as great as in type 2 diabetic individuals of the same age, even though type 1 diabetic individuals usually have fewer additional CVD risk factors. This is likely due to earlier age of onset of diabetes and therefore much longer exposure to hyperglycemia. The incidence of type 1 diabetes is increasing throughout the world. The reasons for this are thought to be environmental although the exact nature of the environmental precipitants is not well understood. In contrast to type 2 diabetes, in which it is clear that aerobic exercise improves glycemic control, studies in type 1 diabetes have generally not found a significant beneficial effect for aerobic exercise on glycemic control, even though there is often reduction in insulin requirements and improved insulin sensitivity. This paradoxical finding may be because individuals with type 1 diabetes are at much higher risk of hypoglycaemia than type 2 and tend to increase their carbohydrate intake in an effort to avoid exercise-induced drops in glucose.

The acute effects of resistance exercise on glycemia in type 1 diabetes have not been established; it is possible that resistance exercise results in a smoother or more predictable decline in blood glucose than aerobic training does, which might reduce fear of hypoglycemia and consequent overcompensation. Resistance exercise training increases insulin receptor protein expression, which is not true of aerobic exercise training .

Study Design: This will be a randomized, controlled trial with a 2 by 2 factorial design (resistance training versus no resistance training; aerobic training versus no aerobic training) in previously inactive subjects with type 1 diabetes. After screening, qualifying subjects will enter a 5-week stabilization/run in period prior to randomization. During this period their diet and insulin therapy will be assessed and optimized, and in weeks 2-5 they will also undergo three supervised sessions of low-intensity exercise per week. Those demonstrating adequate compliance during the run-in period will then be randomized in equal numbers to Aerobic Training (A) progressing to 45 min 3X/wk at 75% of maximum heart rate, Resistance Training (R) 3X/week progressing to 3 sets, 8 repetitions of 8 exercises at the maximum load that can be lifted 8 times (8RM), both Aerobic Training and Resistance Training (AR) or waiting-list control (C). The exercise intervention will take place at YMCAs in metropolitan Ottawa. Subjects cannot be blinded as to group assignment after randomization, but the main study outcomes will be measured by blinded individuals (lab technologists) using objective methods. Subjects randomized to waiting list control will begin a program of their choice (A, R or AR) after all 6-month outcome measures are collected.

Significance: This study addresses questions of clinical and scientific importance. It will help clarify the benefits and risks of aerobic and resistance exercise training in people with type 1 diabetes. Depending on the strength of any differences found, the study will either stand alone or provide pilot data that will set the stage for a larger definitive study. Even if results are substantially different from our expectations, this study will provide valuable new information on the effects of different exercise modalities on metabolic control, body composition, cardiovascular risk factors, and quality of life in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus as defined by the 2003 CDA guidelines (16) requiring insulin therapy starting within one year of diagnosis and continuously thereafter
* Male or female, age 16-45 years, A1c 0.066-0.090
* Physically inactive (see exclusion criteria below)
* Willingness and ability to work closely with the study physicians, nurse and dietitian and follow intensive diabetes therapy including carbohydrate counting, glucose monitoring ≥ 4 times per day, and intensive insulin therapy--either by multiple daily injections (MDI--insulin aspart or lispro before meals and NPH or insulin glargine 1-2X/day) or continuous subcutaneous insulin infusion (CSII) by pump therapy using insulin aspart or lispro for the duration of involvement in the study. CSII will only be an option for those already on CSII prior to entry in the study.

Exclusion Criteria:

* Participation during the previous 4 months in a regular program of exercise or aerobic sports greater than 2 times per week for at least 20 minutes per session, or in any resistance training.
* Hypoglycemia unawareness, or severe hypoglycemia requiring assistance from another person within the previous 3 months.
* "Brittle" diabetes, characterized by frequent and unpredictable hypoglycemia (even if not requiring assistance from others) and hyperglycemia.
* Restrictions in physical activity due to disease: intermittent claudication, severe peripheral neuropathy or active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis.
* Known or suspected clinically significant gastroparesis.
* Body mass index less than or equal to 32 kg/m2.
* Fasting serum c-peptide less than 0.2 nmol/l.
* Recent significant weight change (increase or decrease of 5% of body weight during the two months before enrollment).
* An expected requirement within the subsequent 6 months for medications (other than insulin) that will affect glucose metabolism (e.g. corticosteroids).
* If age < 18 yr, linear growth of 1cm during the previous year.
* Significant renal disease: serum creatinine greater than 200 mEq/l. or proteinuria > 1 g/24 hours.
* Uncontrolled hypertension: BP > 150 mm Hg systolic or > 95 mm Hg diastolic in a sitting position.
* Other illness, judged by the patient or investigators to make participation in this study inadvisable.
* Cognitive deficit resulting in inability to understand or comply with instructions.
* Pregnancy at the start of the study, or intention to become pregnant in the next year.
* Inability to communicate in English or French.
* Unwillingness to sign informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-07; Primary Completion 2010-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
HbA1c at the end of the 6-month exercise period | end of study

SECONDARY OUTCOMES:
frequency of hypoglycemia | end of study
fructosamine | end of study
blood pressure | end of study
lipid concentrations | end of study
apolipoproteins A1 and B | end of study
C-reactive protein | end of study
FFA | end of study
body composition (CT & DEXA) | end of study
compliance with the exercise | end of study
quality of life | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Sigal, Principal Investigator — The Ottawa Health Research Institute, The Ottawa Hospital, The University of Ottawa; Gary Goldfield, Principal Investigator — Children's Hospital of Eastern Ontario; Glen Kenny, Principal Investigator — University of Ottawa; Stasia Hadjiyannakis, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Ottawa Health Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- See also: Related Info — http://www.ohri.ca